CLINICAL TRIAL: NCT06413355
Title: Fibroblast Activating Protein (FAP) PET/CT in Adults With Fibrotic Conditions
Brief Title: FAPI-74 PET/CT in Adults With Fibrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19923; 853610 (Other: UPENN IRB)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Fibrosis (Morphologic Abnormality)
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FAPI-74 PET/CT Scan (Experimental): Head and neck cancer (up to 15 subjects), post tubercular lung disease (PTLD, up to 10 subjects), Cardiac Sarcoidosis and Exploratory (up to 10 subjects each) with fibrosis-inducing medical conditions that are known or suspected to cause tissue fibrosis (e.g. cancer-associated, postinfection, post-radiation, pre/post-transplant, cardiac, liver, kidney or pulmonary fibrosis).
  Interventions: Drug: [F-18]-FAPI-74

INTERVENTIONS:
Drug: [F-18]-FAPI-74 — A positron-emitting radiopharmaceutical that has been studied in animals for selective measurement of the in vivo expression of FAP with positron emission tomography (PET/CT).
  Other Names: [18F] aluminium fluorine ((S)-2,2'(7- (2-(4-(3-(4-(2-(2- cyanopyrrolidin-1-yl)-2 oxoethylcarbamoyl)quinolin-6-yloxy) propyl)piperazin-1-yl)-2-oxoethyl)-1,4,7- triazonane-1,4-diyl)diacetic acid

SUMMARY:
This protocol is intended as a basket protocol designed to evaluate the use of Fibroblast Activating Protein (FAP) PET/CT in imaging the presence of fibrosis caused by a variety of medical conditions where fibrosis is believed to lead to pathological effects and poor prognosis.

DETAILED DESCRIPTION:
A study to evaluate subjects with fibrosis-inducing medical conditions that are known or suspected to cause tissue fibrosis (e.g. cancer-associated, post-infection, post-radiation, pre or post-transplant, cardiac, liver, kidney or pulmonary fibrosis). This protocol is intended to expand as needed with imaging arms designed to evaluate the use of Fibroblast Activating Protein (FAP) PET/ CT in imaging the presence fibrosis caused by medical conditions where fibrosis is believed to lead to pathological effects and poor prognosis.

[18F]-FAPI-74 is a positron emitting radiolabeled FAP inhibitor that will be used with a positron emission tomography/computed tomography (PET/CT) scan that will be completed in each subject who has a clinical suspicion of fibrotic disease.

PET/CT imaging will be used to evaluate the distribution of fibroblast activating protein (FAP) in major organs and other tissues affected with fibrotic diseases or conditions. This is an observational study in that [F-18]-FAPI-74 PET/CT will not be used to direct treatment decisions. While patients and referring physicians will not be blinded to the [F-18]-FAPI-74 PET/CT results, any medical or treatment decisions related to their underlying clinical diagnosis will be made by the treating physicians based upon clinical criteria.

After injection of [F-18]-FAPI-74, patients will undergo a vertex to mid-thigh scan, starting at approximately 15 minutes post injection. PET/CT imaging sessions will include an injection of approximately 8.0 mCi (expected range of doses is expected to be 6.0-8.0 mCi) of [F-18]-FAPI-74 intravenously. Data will be collected to evaluate uptake of [F-18]-FAPI-74 in sites of suspected fibrosis and in major organs.

An optional second PET/CT using [F-18]-FAPI-74 can be considered at the request of the investigators at any clinically relevant time point for the H&N, Exploratory and Cardiac Sarcoidosis cohorts. This second scan may be used to quantify the changes in fibrosis over time as part of the natural progression of the fibrotic condition, or to observe changes in [F-18]-FAPI-74 uptake in response to therapeutic interventions.

Imaging cohorts include:

Head and neck cancer (up to 15 patients) Post tubercular lung disease (PTLD, up to 10 patients) Cardiac Sarcoidosis (up to 10 patients) Exploratory Cohort (Pilot studies for generating clinical data to support use of the radiotracer for FAP targeted therapies, up to 10 patients)

Uptake of [F-18]-FAPI-74 may be compared to other clinical pathology or lab results related to the presence of fibrosis (e.g. tissue sequencing, genomics, immunohistochemistry, ELISA, and similar assays))

ELIGIBILITY:
Inclusion Criteria (by cohort)

Head and Neck Cancer Cohort:

1. Participants will be ≥ 21 years of age
2. Diagnosis of oropharyngeal squamous cell carcinoma (OPSCC)
3. Determined to be surgical candidates
4. History of known or suspected fibrosis-inducing medical condition

PTLD Cohort:

1. Participants will be ≥ 21 years of age
2. Diagnosed with microbiologically confirmed DS-pTB (culture or PCR positive)
3. History of known or suspected fibrosis-inducing medical condition.
4. Patient-reported completion of TB treatment within 2 years of enrollment.

Cardiac Sarcoidosis Cohort:

1. Participants will be ≥ 21 years of age
2. FDG PET/CT scan consistent with metabolically active cardiac sarcoidosis
3. Clinical suspicion of cardiac involvement defined as the presence of any of the following:

   1. High degree A-V nodal block
   2. Reduced left or right ventricular systolic fusion
   3. History of ventricular arrhythmias
   4. Unexplained syncope

Exploratory Cohort:

1. Participants will be ≥ 21 years of age
2. History of known or suspected fibrosis-inducing medical condition.

All Cohorts:

1. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria (by cohort)

Head and Neck Cancer Cohort:

1. Patient is not eligible for tissue resection

PTLD Cohort:

1. Diagnosed with TB that is resistant to rifampin per medical record review
2. History of alternative pulmonary disease per medical record review or patient self-report
3. Have been administered corticosteroids or any other systemic investigational agents within 3 months of screening per medical record review or patient self-report
4. Have symptoms or signs suggestive of active TB at the time of pre-screening per patient self-report

All Cohorts:

1. Women of childbearing potential may not be pregnant or breast-feeding. A negative pregnancy test will be required before [F-18]-FAPI-74injection.
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
3. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study
4. Treatment with a therapeutic agent targeting fibroblast activation protein (FAP) within 1 month prior to study enrollment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Overall FAPI-74 PET/CT Image Analysis | 3 years
  The overall quality of the generated images will be evaluated. Initial imaging of the vertex to mid-thigh will be used to investigate regional tracer uptake in suspected sites of fibrosis and normal tissues for this novel radiotracer. Uptake and retention of [F-18]-FAPI-74 in known or suspected sites of fibrotic disease will be evaluated visually by trained radiology readers, the principal investigator, or designee. A number of analysis methods may be tested to identify the optimal method for analyses for future studies with this radiotracer. [F-18]-FAPI-74 PET/CT scans will be interpreted both qualitatively and quantitatively.
Head and Neck Cancer FAPI-74 PET/CT Image Analysis | 3 years
  [18F]-FAPi74 PET/CT data: Areas of uptake in tumors and healthy tissue will be measured by SUVmax and semiquantitative analysis will be conducted. In each case, lesion uptake will be marked as low, medium, and high avidity. Each lesion and lymph node will be separately measured and quantified. Measurements will be made by Dr. Sellmyer and co-Investigators (n=3).
PTLD FAPI-74 PET/CT Image Analysis | 3 years
  Quantitative interpretation of FAP expression, will be recorded as a Standardized Uptake Value (SUV). Max, mean, and peak SUV values will be recorded for a region-of-interest encompassing a single primary lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Sellmyer, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No